CLINICAL TRIAL: NCT00795951
Title: Clinical Evaluation of T.R.U.E. TEST® Panel 1.1, 2.1 and 3.1: in Children and Adolescents
Brief Title: Clinical Evaluation of T.R.U.E. TEST in Children and Adolescents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allerderm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MEKOS 07 29P1/2/3/401
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2013-12

CONDITIONS: Dermatitis, Contact
Keywords: allergic; contact dermatitis; contact allergy; Type IV; Children; TRUE TEST
MeSH Terms: conditions — Dermatitis, Contact; Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRUE Test panels 1.1, 2.1, 3.1 (Experimental): All subjects were patched with 3 T.R.U.E. Test panels containing 28 allergens and 1 negative control.
  Interventions: Biological: T.R.U.E. Test

INTERVENTIONS:
Biological: T.R.U.E. Test — 48 hour application of 28 allergens and negative control
  Other Names: NA no other names

SUMMARY:
Open, prospective, single-site, non-randomized study of the efficacy and safety of T.R.U.E. TEST allergens in children and adolescents ages 6-18.

DETAILED DESCRIPTION:
Three T.R.U.E. TEST panels (1.1, 2.1 and 3.1) containing 28 allergens and a negative control will be applied to the skin on the subject's back and worn for approximately 48 hours. Patch test site skin reactions will be evaluated at days 2, 3 (+1), 7 and 21 following panel application

ELIGIBILITY:
Inclusion Criteria:

* Symptoms and history potentially consistent with allergic contact dermatitis based on symptoms and clinical history (i.e., subjects are visiting the clinic/physician to diagnose, treat or resolve this condition).
* Children and adolescents 6 to 18 years of age, and in general good health.
* Adolescent females 15 years of age or older (or with menarche) must consent to a urine pregnancy test; urine test results must be negative for study inclusion.
* Informed consent must be signed and understood by subject. If underage, informed consent must be signed and understood by parent or legal guardian, consistent with all institutional, local and national regulations.

Exclusion Criteria:

* Topical corticosteroid treatment during the last 7 days on or near the test area.
* Systemic treatment with corticosteroids or other immunosuppressive during the last 7 days.
* Subjects currently receiving (or received during the previous 3 weeks) other investigational drugs, treatments or devices, or participating in another clinical study.
* Treatment with ultraviolet (UV) light (including tanning) during the previous 3 weeks.
* Acute dermatitis outbreak or dermatitis on or near the test area on the back.
* Subjects unable to comply with activity restrictions (e.g., protecting test panels from excess moisture due to showering or vigorous activity).
* Subjects unable or unwilling to comply with multiple return visits.
* Female subjects 15 years of age (or with onset of menarche) and older unable to consent to a urine pregnancy test, or those with a positive pregnancy test.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 102 (Actual)
Dates: Start 2008-11; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Eichenfield, MD, Principal Investigator — UCSD School of Medicine
Locations (1):
- Rady Children's Hospital, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Single Site- Rady Children's Hospital Recruiting Period-09 December 2008 (first subject enrolled) 27 October 2009 (last subject exited)
Pre-assignment Details: No significant events or approaches
Groups:
- All Subjects: T.R.U.E. Test Allergen Panel evaluations
Period: Overall Study
Arm/Group | All Subjects
Started | 102
Completed | 100
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Single Arm Study: All subjects were patched with TRUE Test panels 1.1, 2.1 and 3.1
Arm/Group | Single Arm Study
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 102
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 49
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Positive Reactions: Nickel Sulfate
Description: Number of subjects with positive reactions (score of 1+, 2+ or 3+) at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 30

2. Primary Outcome: Positive Reactions: Neomycin Sulfate
Description: Number of subjects with positive reactions (score of 1+, 2+ or 3+) at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 8

3. Primary Outcome: Positive Reactions: Wool Alcohol
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 16

4. Primary Outcome: Positive Reactions: Potassium Dichromate
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 9

5. Primary Outcome: Positive Reactions: Caine Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 72-96 hours after patch application, Visit 4: 1 week after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Groups:
- Diagnostic Performance: T.R.U.E. Test allergen panel evaluations
Arm/Group | Diagnostic Performance
Number analyzed (Participants) | 100
participants | 0

6. Primary Outcome: Positive Reactions: Fragrance Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 13

7. Primary Outcome: Positive Reactions: Colophony
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 9

8. Primary Outcome: Positive Reactions: Paraben Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

9. Primary Outcome: Positive Reactions: Negative Control
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4.
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

10. Primary Outcome: Positive Reactions: Balsam of Peru
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 11

11. Primary Outcome: Positive Reactions: Ethylenediamine Dihydrochloride
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days week after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 5

12. Primary Outcome: Positive Reactions: Cobalt Dichloride
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 13

13. Primary Outcome: Positive Reactions: P-tert Butylphenol Formadehyde Resin
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 17

14. Primary Outcome: Positive Reactions: Epoxy Resin
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 4

15. Primary Outcome: Positive Reactions: Carba Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 7

16. Primary Outcome: Positive Reactions: Black Rubber Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

17. Primary Outcome: Positive Reactions: Cl+Me-Isothiazolinone
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 4

18. Primary Outcome: Positive Reactions: Quaternium-15
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 4

19. Primary Outcome: Positive Reactions: Mercaptobenzothiazole
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

20. Primary Outcome: Positive Reactions: p-Phenylenediamine
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

21. Primary Outcome: Positive Reactions: Formaldehyde
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 7

22. Primary Outcome: Positive Reactions: Mercapto Mix
Description: Number of subjects with positive reactions at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

23. Primary Outcome: Positive Reactions: Thimerosal
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 4

24. Primary Outcome: Positive Reactions: Thiuram Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 7

25. Primary Outcome: Positive Reactions: Diazolidinyl Urea
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 5

26. Primary Outcome: Positive Reactions: Imidazolidinyl Urea
Description: Number of subjects with positive reactions at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

27. Primary Outcome: Positive Reactions: Budesonide
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

28. Primary Outcome: Positive Reactions: Tixocortol-21-pivalate
Description: Number of subjects with positive reactions at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 8

29. Primary Outcome: Positive Reactions: Quinoline Mix
Description: Number of subjects with positive reactions recorded at visit 3 and/or visit 4
Time Frame: Visit 3: 3-4 days after patch application, Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

30. Secondary Outcome: Late Reactions: Nickel Sulfate
Description: Number of subjects with late reactions, defined as a positive reaction that initially occurs at day 7 (visit 4) or later.
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

31. Secondary Outcome: Late Reactions: Neomycin Sulfate
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

32. Secondary Outcome: Late Reactions: Wool Alcohol
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

33. Secondary Outcome: Late Reactions: Potassium Dichromate
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

34. Secondary Outcome: Late Reactions: Caine Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | Diagnostic Performance
Number analyzed (Participants) | 100
participants | 0

35. Secondary Outcome: Late Reactions: Fragrance Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

36. Secondary Outcome: Late Reactions: Colophony
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

37. Secondary Outcome: Late Reactions: Paraben Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

38. Secondary Outcome: Late Reactions: Negative Control
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

39. Secondary Outcome: Late Reactions: Balsam of Peru
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

40. Secondary Outcome: Late Reactions: Ethylenediamine Dihydrochloride
Description: as for outcome 30
Time Frame: Visit 4: 7 days week after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

41. Secondary Outcome: Late Reactions: Cobalt Dichloride
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

42. Secondary Outcome: Late Reactions: P-tert Butylphenol Formadehyde Resin
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

43. Secondary Outcome: Late Reactions: Epoxy Resin
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

44. Secondary Outcome: Late Reactions: Carba Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

45. Secondary Outcome: Late Reactions: Black Rubber Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

46. Secondary Outcome: Late Reactions: Cl+Me-Isothiazolinone
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

47. Secondary Outcome: Late Reactions: Quaternium-15
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

48. Secondary Outcome: Late Reactions: Mercaptobenzothiazole
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

49. Secondary Outcome: Late Reactions: p-Phenylenediamine
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

50. Secondary Outcome: Late Reactions: Formaldehyde
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

51. Secondary Outcome: Late Reactions: Mercapto Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

52. Secondary Outcome: Late Reactions: Thimerosal
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

53. Secondary Outcome: Late Reactions: Thiuram Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

54. Secondary Outcome: Late Reactions: Diazolidinyl Urea
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

55. Secondary Outcome: Late Reactions: Imidazolidinyl Urea
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

56. Secondary Outcome: Late Reactions: Budesonide
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

57. Secondary Outcome: Late Reactions: Tixocortol-21-pivalate
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

58. Secondary Outcome: Late Reactions: Quinoline Mix
Description: as for outcome 30
Time Frame: Visit 4: 7 days after patch application or Visit 5: 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

59. Secondary Outcome: Persistent Reactions: Nickel Sulfate
Description: Number of subjects with persistent reactions defined as positive reactions identified at visit 3 or 4 that are still present at the next visit.
Time Frame: Visit 3: 3-4 days after patch application through Visit 4: 7 days after patch application and/or Visit 5 21 days after patch application
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 16

60. Secondary Outcome: Persistent Reactions: Neomycin Sulfate
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 5

61. Secondary Outcome: Persistent Reactions: Wool Alcohol
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 6

62. Secondary Outcome: Persistent Reactions: Potassium Dichromate
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 3

63. Secondary Outcome: Persistent Reactions: Caine Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

64. Secondary Outcome: Persistent Reactions: Fragrance Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 5

65. Secondary Outcome: Persistent Reactions: Colophony
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 4

66. Secondary Outcome: Persistent Reactions: Paraben Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

67. Secondary Outcome: Persistent Reactions: Negative Control
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

68. Secondary Outcome: Persistent Reactions: Balsam of Peru
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

69. Secondary Outcome: Persistent Reactions: Ethylenediamine Dihydrochloride
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 4

70. Secondary Outcome: Persistent Reactions: Cobalt Dichloride
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 5

71. Secondary Outcome: Persistent Reactions: P-tert Butylphenol Formadehyde Resin
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 6

72. Secondary Outcome: Persistent Reactions: Epoxy Resin
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

73. Secondary Outcome: Persistent Reactions: Carba Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

74. Secondary Outcome: Persistent Reactions: Black Rubber Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

75. Secondary Outcome: Persistent Reactions: Cl+Me-Isothiazolinone
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 3

76. Secondary Outcome: Persistent Reactions: Quaternium-15
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

77. Secondary Outcome: Persistent Reactions: p-Phenylenediamine
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

78. Secondary Outcome: Persistent Reactions: Formaldehyde
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

79. Secondary Outcome: Persistent Reactions: Mercapto Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

80. Secondary Outcome: Persistent Reactions: Thimerosal
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

81. Secondary Outcome: Persistent Reactions: Thiuram Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

82. Secondary Outcome: Persistent Reactions: Diazolidinyl Urea
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 2

83. Secondary Outcome: Persistent Reactions: Imidazolidinyl Urea
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

84. Secondary Outcome: Persistent Reactions: Budesonide
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

85. Secondary Outcome: Persistent Reactions: Tixocortol-21-pivalate
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 3

86. Secondary Outcome: Persistent Reactions: Quinoline Mix
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 0

87. Secondary Outcome: Persistent Reactions: Mercaptobenzothiazole
Description: as for outcome 59
Time Frame: as for outcome 59
Population: Number of participants analyzed includes all subjects who completed the study.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
participants | 1

88. Secondary Outcome: Panel Adhesion Evaluation
Description: Panel Adhesion was evaluated according to the following score scale: Off: Test panel fell off, Poor: little to no skin to panel contact, Fair: skin to panel contact variable, tape edges lifting, Good: skin contact acceptable, some tape edges loose; Excellent, skin contact good, tape edges adherent.
Time Frame: Visit 2 (day 1) prior to panel removal.
Population: All subjects who completed the study are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
Participants
  Panel 1 Adhesion Scores: Excellent | 71
  Panel 1 Adhesion Scores: Good | 19
  Panel 1 Adhesion Scores: Fair | 8
  Panel 1 Adhesion Scores: Poor | 2
  Panel 1 Adhesion Scores: Fell off | 0
  Panel 2 Adhesion Scores: Excellent | 72
  Panel 2 Adhesion Scores: Good | 19
  Panel 2 Adhesion Scores: Fair | 9
  Panel 2 Adhesion Scores: Poor | 0
  Panel 2 Adhesion Scores: Fell off | 0
  Panel 3 Adhesion Scores: Excellent | 82
  Panel 3 Adhesion Scores: Good | 14
  Panel 3 Adhesion Scores: Fair | 3
  Panel 3 Adhesion Scores: Poor | 1
  Panel 3 Adhesion Scores: Fell off | 0

89. Secondary Outcome: Panel Irritation
Description: Panel Irritation was scored according to the following descriptors; None, Weak, Moderate, Strong (not defined in protocol)
Time Frame: Visit 2 (day 1) following to panel removal.
Population: All subjects who completed the study are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
Participants
  Panel 1 Irritation: None | 38
  Panel 1 Irritation: Weak | 43
  Panel 1 Irritation: Moderate | 16
  Panel 1 Irritation: Strong | 3
  Panel 2 Irritation: None | 37
  Panel 2 Irritation: Weak | 43
  Panel 2 Irritation: Moderate | 16
  Panel 2 Irritation: Strong | 4
  Panel 3 Irritation: None | 40
  Panel 3 Irritation: Weak | 40
  Panel 3 Irritation: Moderate | 18
  Panel 3 Irritation: Strong | 2

90. Secondary Outcome: Subject Reported Itching and Burning
Description: Subject reported itching/burning was scored according to the following descriptors; None, Weak, Moderate, Strong (not defined in protocol)
Time Frame: Visit 2 (day 1) following to panel removal.
Population: All subjects who completed the study are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | All Subjects
Number analyzed (Participants) | 100
Participants
  Panel 1 Itching and Burning: None | 33
  Panel 1 Itching and Burning: Weak | 34
  Panel 1 Itching and Burning: Moderate | 12
  Panel 1 Itching and Burning: Strong | 21
  Panel 2 Itching and Burning: None | 44
  Panel 2 Itching and Burning: Weak | 32
  Panel 2 Itching and Burning: Moderate | 15
  Panel 2 Itching and Burning: Strong | 9
  Panel 3 Itching and Burning: None | 60
  Panel 3 Itching and Burning: Weak | 23
  Panel 3 Itching and Burning: Moderate | 5
  Panel 3 Itching and Burning: Strong | 12

ADVERSE EVENTS:
Time Frame: The Adverse Event-Reporting Period for each study subject began at application of the patch test and ended with the Day 21 visit.
Groups:
- Safety: Adverse Events
Arm/Group | Safety
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 42/102
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety (N=102)
Worsening of rash (Skin and subcutaneous tissue disorders) | 26 (34)
Flare-up of rash (Skin and subcutaneous tissue disorders) | 2 (2)
Boil on forehead (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Headache (Vascular disorders) | 2 (2)
Fever (Infections and infestations) | 2 (2)
Reaction around panel 2.1 (Skin and subcutaneous tissue disorders) | 1 (1)
Edema, vesiculation pain on hands (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening of underlying condition (Skin and subcutaneous tissue disorders) | 1 (1)
Slight worsening of spot on leg (Skin and subcutaneous tissue disorders) | 1 (1)
Lesion on right thumb (Skin and subcutaneous tissue disorders) | 1 (1)
Worsening of dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Reaction on place of panel (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No